CLINICAL TRIAL: NCT01287286
Title: Cancers Treated With Combination of Antrodia Cinnamomea and Chemotherapy- a Double Blinded, Randomized, Placebo-controlled Trial
Brief Title: Cancers Treated With Combination of Antrodia Cinnamomea and Chemotherapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: New Bellus Enterprises (Unknown)
Responsible Party: Yu-Chiang Hung / MD, PhD, Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital- Kaohsiung Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: XMRPG890251
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-01

CONDITIONS: Neoplasm; Functional Gastrointestinal Disorder
Keywords: Cancers; Antrodia cinnamomea; Chemotherapy; Gastrointestinal Disorder
MeSH Terms: conditions — Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-Can (Experimental): Antrodia cinnamomea and concomitant chemotherapy
  Interventions: Dietary Supplement: AC-Can
- control (Placebo Comparator): Placebo and concomitant chemotherapy
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: AC-Can — Antrodia cinnamomea compounds of 15 milliliters liquid per pack, oral post meal, twice in a day for 30 days
  Other Names: AC
  Arms: AC-Can
Dietary Supplement: placebo — Placebo of 15 milliliters liquid per pack, oral post meal, twice in a day for 30 days
  Arms: control

SUMMARY:
The purpose of this study is to investigate if food supplements,Antrodia cinnamomea, could minimize the gastrointestinal symptom of cancer patients with chemotherapy.

DETAILED DESCRIPTION:
In our unpublished report shows that patients who took Antrodia Cinnamomea compound of 15 milliliters liquid twice in a day, might help white blood cells, red blood cells and hemoglobin increase after 2 months; liver glutamic pyruvic transaminase(GPT) index mitigation, P <0.05 difference statistically; In addition, liver glutamate oxaloacetate transaminase(GOT) and biochemical index of renal function had no abnormal data statistically. However, cancer patients with gastrointestinal disorders after chemotherapy is known to be a common side effect, we seek to investigate if Antrodia Cinnamomea improves the function of gastrointestinal system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Cancer.
* Age ≦ 80 years old and ≧ 18 years old.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0-2.
* Adequate organ function, including followings Hepatic： Total bilirubin level ≦1.5 x UNL, GOT and GPT ≦ 2.5 x UNL if no liver metastasis; GOT and GPT ≦ 5 x UNL if liver metastasis. Renal： Creatinine level< 1.5 milligram per deciliter or Estimated creatinine clearance(CCr) ≧ 60 milliliter per minute (CCr is estimated by Cockcroft-Gault formula, as appendix II)
* Estimated life expectancy of at least 12 weeks.
* Written(signed) Informed Consent
* Ever treated and poor tolerance with platinum-based or anthracycline- based regimen, likely nausea and vomiting.

Exclusion Criteria:

* Prior participation in any investigational drug study within 28 days
* Active uncontrolled infections or human immunodeficiency virus(HIV) infection
* Significant concurrent medical diseases, such as congestive heart failure, unstable angina, acute or recent myocardial infarction( 6 months before randomization), chronic obstructive pulmonary disease with frequent exacerbation, chronic renal diseases (estimated CCr 60 milliliter per minute), uncontrolled diabetes, uncontrolled hypertension, recent cerebrovascular disease episode( 6 months before randomization )
* With clinically significant Gastrointestinal disorder (e.g. bleeding, inflammation, obstruction or diarrhea)
* Psychiatric disorders that would compromise the patient's compliance or decision.
* Pregnancy or breast feeding.
* Known hypersensitivity to the component of investigational drugs.
* Known or suspected Gilbert's syndrome
* Poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms in case group reduces 10% than control group during chemotherapy. | 1 month
  Post-chemotherapy nausea, vomiting and epigastragia, etc. including gastrointestinal symptom/sign without mention above.

SECONDARY OUTCOMES:
Life quality estimates of 10% improvement than control group. | 3 months
  Life science related questionnairs visit 4 times just before treatment, after intervention 7 days, 30 days and 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chiang Hung, MD, PhD, Principal Investigator — Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital - Kaohsiung Medical Center
Locations (1):
- Division of Haematology and Oncology, Department of Internal Medicine and Traditional Chinese Medicine, Chang Gung Memorial Hospital - Kaohsiung Medical Center, Niaosong, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Tsai MY, Hung YC, Chen YH, Chen YH, Huang YC, Kao CW, Su YL, Chiu HH, Rau KM. A preliminary randomised controlled study of short-term Antrodia cinnamomea treatment combined with chemotherapy for patients with advanced cancer. BMC Complement Altern Med. 2016 Aug 26;16(1):322. doi: 10.1186/s12906-016-1312-9. PMID 27565426